CLINICAL TRIAL: NCT03453281
Title: Central Macular Thickness, Macular Electroretinogram, and Visual Acuity in Patients With Diabetic Macular Edema After Intravitreal Aflibercept Injection. A One Month Pre-Post Intervention Follow Up Study
Brief Title: Early Anatomical, Physiological, and Clinical Changes in Diabetic Macular Edema After Intravitreal Aflibercept Injection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Martin Hertanto, Resident, Dept. of Ophthalmology, Faculty of Medicine Universitas Indonesia, Indonesia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-07-0750
Record Dates: First submitted 2018-02-26; First posted 2018-03-05 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Diabetic Macular Edema; Diabetic Retinopathy; Clinically Significant Macular Edema
Keywords: Aflibercept; Diabetic Macular Edema; Electroretinogram; Central Macular Thickness; ETDRS
MeSH Terms: conditions — Diabetic Retinopathy | interventions — aflibercept

STUDY DESIGN:
Intervention Model Description: Every subject was given the same treatment (intravitreal Aflibercept injection).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Aflibercept Injection [Eylea] (Experimental): Intravitreal injection of 2 mg in 0.05 ml Aflibercept. Frequency: once Duration: 10-15 minutes
  Interventions: Drug: Aflibercept Injection [Eylea]

INTERVENTIONS:
Drug: Aflibercept Injection [Eylea] — Intravitreal Aflibercept injections were performed by vitreoretinal consultant at the place of study.
  Other Names: Intravitreal Aflibercept injection; Intravitreal Eylea injection; Intravitreal anti VEGF injection; Aflibercept intravitreal injection; Eylea intravitreal injection; Anti VEGF intravitreal injection

SUMMARY:
This is a one month pre post intervention study. Subjects with diabetic macular edema were given intravitreal anti VEGF (Aflibercept) injection. Central retinal thickness, macular electrophysiology, and visual acuity were observed one week and one month after injection was given to the eye to describe early anatomical, physiological, and clinical changes. We hypothesized that changes to these outcomes can be found and documented.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 y.o.
* Diagnosed with Type 1 or 2 Diabetes Mellitus
* Have either one of mild non-proliferative diabetic retinopathy (NPDR), moderate NPDR, severe NPDR, or Proliferative Diabetic Retinopathy with clinically significant macular edema according to Early Treatment for Diabetic Retinopathy Study (ETDRS) criteria
* Best corrected visual acuity between one meter finger counting to 6/12 (ETDRS chart)
* Minimum Central Macular Thickness by Optical Coherence Tomography examination of 250 um
* Willing to participate and sign the informed consent.

Exclusion Criteria:

* Ongoing pregnancy or planning to be pregnant for the next 6 months.
* Media opacity (e.g. corneal scar, corneal edema, cataract, vitreous hemorrhage) which make macular OCT not possible
* History of intraocular surgery in the last 6 months
* Vitreoretinal surface disorders e.g. epiretinal membrane, vitreoretinal traction
* History of panretinal laser photocoagulation in the last 6 months
* Presence of iris neovascularization
* History of eye trauma
* HbA1c level > 10,0 %
* Any other contraindication(s) for intravitreal anti VEGF injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-05-18 (Actual)

PRIMARY OUTCOMES:
Central macular thickness | One month after intravitreal Aflibercept injection
  Central macular thickness (CMT) measured by Cirrus® HD OCT, Carl Zeiss, Germany [in µm]

SECONDARY OUTCOMES:
Central macular thickness | One week after intravitreal Aflibercept injection
  Central macular thickness (CMT) measured by Cirrus® HD OCT, Carl Zeiss, Germany [in µm]
Amplitude of P1 wave | One week after intravitreal Aflibercept injection
  Amplitude of P1 wave in multifocal electroretinogram (MfERG) measured by Electroretinography (Vision Monitor MonPackONE, Metrovision, France) [in nV/deg2]
Amplitude of P1 wave | One month after intravitreal Aflibercept injection
  Amplitude of P1 wave in multifocal electroretinogram (MfERG) measured by Electroretinography (Vision Monitor MonPackONE, Metrovision, France) [in nV/deg2]
Amplitude of N1 wave | One week after intravitreal Aflibercept injection
  Amplitude of N1 wave in MfERG measured by Electroretinography (Vision Monitor Monpack one, Metrovision, France) [in nV/deg2]
Amplitude of N1 wave | One month after intravitreal Aflibercept injection
  Amplitude of N1 wave in MfERG measured by Electroretinography (Vision Monitor Monpack one, Metrovision, France) [in nV/deg2]
Amplitude of N2 wave | One week after intravitreal Aflibercept injection
  Amplitude of N2 wave in MfERG measured by Electroretinography (Vision Monitor Monpack one, Metrovision, France) [in nV/deg2]
Amplitude of N2 wave | One month after intravitreal Aflibercept injection
  Amplitude of N2 wave in MfERG measured by Electroretinography (Vision Monitor Monpack one, Metrovision, France) [in nV/deg2]
Implisit time of P1 wave | One week after intravitreal Aflibercept injection
  Implisit time of P1 wave in MfERG measured by Electroretinography (Vision Monitor Monpack one, Metrovision, France) [in nV/deg2]
Implisit time of P1 wave | One month after intravitreal Aflibercept injection
  Implisit time of P1 wave in MfERG measured by Electroretinography (Vision Monitor Monpack one, Metrovision, France) [in nV/deg2]
Implisit time of N1 wave | One week after intravitreal Aflibercept injection
  Implisit time of N1 wave in MfERG measured by Electroretinography (Vision Monitor Monpack one, Metrovision, France) [in nV/deg2]
Implisit time of N1 wave | One month after intravitreal Aflibercept injection
  Implisit time of N1 wave in MfERG measured by Electroretinography (Vision Monitor Monpack one, Metrovision, France) [in nV/deg2]
Implisit time of N2 wave | One week after intravitreal Aflibercept injection
  Implisit time of N2 wave in MfERG measured by Electroretinography (Vision Monitor Monpack one, Metrovision, France) [in nV/deg2]
Implisit time of N2 wave | One month after intravitreal Aflibercept injection
  Implisit time of N2 wave in MfERG measured by Electroretinography (Vision Monitor Monpack one, Metrovision, France) [in nV/deg2]
Best corrected visual acuity | One week after intravitreal Aflibercept injection
  Best corrected visual acuity (BCVA) measured by ETDRS chart [in LogMAR]
Best corrected visual acuity | One month after intravitreal Aflibercept injection
  Best corrected visual acuity (BCVA) measured by ETDRS chart [in LogMAR]
Best corrected visual acuity (number of letters) | One week after intravitreal Aflibercept injection
  BCVA (number of letters) measured by ETDRS chart [in number of letters]
Best corrected visual acuity (number of letters) | One month after intravitreal Aflibercept injection
  BCVA (number of letters) measured by ETDRS chart [in number of letters]
Uncorrected visual acuity | One week after intravitreal Aflibercept injection
  Uncorrected visual acuity (UCVA) measured by ETDRS chart [in LogMAR]
Uncorrected visual acuity | One month after intravitreal Aflibercept injection
  Uncorrected visual acuity (UCVA) measured by ETDRS chart [in LogMAR]
Uncorrected visual acuity (number of letters) | One week after intravitreal Aflibercept injection
  UCVA (number of letters) measured by ETDRS chart [in number of letters]
Uncorrected visual acuity (number of letters) | One month after intravitreal Aflibercept injection
  UCVA (number of letters) measured by ETDRS chart [in number of letters]

CONTACTS AND LOCATIONS:
Overall Officials: Anggun Yudantha, dr., SpM(K), Principal Investigator — Dept. of Ophthalmology, Faculty of Medicine Universitas Indonesia, RSCM Kirana; Syntia Nusanti, dr., SpM(K), Principal Investigator — Dept. of Ophthalmology, Faculty of Medicine Universitas Indonesia, RSCM Kirana
Locations (1):
- Dept. of Ophthalmology, Faculty of Medicine Universitas Indonesia, RSCM Kirana, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided
The data obtained in this study belong not only to the investigator, but also partly to the institution where this study is conducted. Any request regarding participant data will be considered and permissions will be granted when all the stakeholders approved.